CLINICAL TRIAL: NCT06831604
Title: Ultrasound Guided Superficial Cervical Plexus Block With Either Clavipectoral Fascial Plane Block or Interscalene Brachial Block for Clavicle Surgeries Anesthesia: A Randomized Controlled Trial
Brief Title: Superficial Cervical Plexus Block With Either Clavipectoral Fascial Plane Block or Interscalene Brachial Block for Clavicle Surgeries Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Aboeldahab, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36265MD331/12/24
Record Dates: First submitted 2025-02-08; First posted 2025-02-18 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Ultrasound; Superficial Cervical Plexus Block; Clavipectoral Fascial Plane Block; Interscalene Brachial Block; Clavicle Surgeries
MeSH Terms: interventions — small cardioactive peptide B

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Patients will receive Superficial Cervical Plexus Block (SCPB) and Clavipectoral Fascial Plane Block (CPB).
  Interventions: Drug: Superficial Cervical Plexus Block (SCPB) and Clavipectoral Fascial Plane Block (CPB)
- Group II (Experimental): Patients will receive Superficial Cervical Plexus Block (SCPB) and Interscalene Brachial Block (ISBP).
  Interventions: Drug: Superficial Cervical Plexus Block (SCPB) and Interscalene Brachial Block (ISBP)

INTERVENTIONS:
Drug: Superficial Cervical Plexus Block (SCPB) and Clavipectoral Fascial Plane Block (CPB) — Patients will receive Superficial Cervical Plexus Block (SCPB) and Clavipectoral Fascial Plane Block (CPB).
  Other Names: Group I
  Arms: Group I
Drug: Superficial Cervical Plexus Block (SCPB) and Interscalene Brachial Block (ISBP) — Patients will receive Superficial Cervical Plexus Block (SCPB) and Interscalene Brachial Block (ISBP)
  Other Names: Group II
  Arms: Group II

SUMMARY:
This study aims to evaluate and compare the efficacy and safety of ultrasound guided superficial cervical plexus block (SCPB) with either clavipectoral fascial plane block (CPB) or interscalene brachial plexus block (ISBP) as an anesthetic technique for clavicle surgeries.

DETAILED DESCRIPTION:
Clavicular fracture is the most common injury in the shoulder, it occurs in 35% of shoulder girdle fractures. Clavicle surgeries often involve addressing fractures, dislocations, or corrective procedures, and they generally require precise and effective pain control.

Traditional superficial cervical plexus block (SCPB) combined with interscalene brachial plexus block (ISBP) can be used in the operation of clavicle fracture.

The SCPB targets the cervical plexus, providing sensory anesthesia to the skin overlying the cervical and upper thoracic regions. It is often used in conjunction with other blocks to enhance analgesia in the upper shoulder and clavicle area.

The ISBP block involves the administration of local anesthetic at the level of the brachial plexus, typically performed between the anterior and middle scalene muscles. This approach provides comprehensive analgesia for the shoulder, upper arm, and part of the clavicular area.

Clavipectoral fascial plane block (CPB) is a new regional nerve block and can be used in anesthesia and postoperative analgesia for clavicle fracture surgery. CPB provides analgesia to the clavicular region and the upper shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I, II.
* Patients with unilateral clavicular fractures undergo elective internal fixation of clavicle fractures.

Exclusion Criteria:

* Coagulopathy.
* Patients with infection at block site.
* Allergy to local anesthetics.
* Patient with morbid obesity (body mass index >35 kg/m2).
* Pre-existing neurological disease.
* Difficult communication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Success rate | Intraoperatively
  The block will be considered successful when complete sensory block is achieved within 45 min after injection of the study drug and inadequate block will be converted to general anesthesia and excluded from the study.

SECONDARY OUTCOMES:
First request of the rescue analgesia | 24 hours postoperatively
  First request of the rescue analgesia will be recorded from the end of surgery till first dose of morphine administrated
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 2 mg bolus if the visual Analogue Scale (VAS)> 3 to be repeated after 30 min if pain persists until the VAS < 4. Each patient will be instructed about postoperative pain assessment with VAS. VAS (0 represents "no pain" while 10 represents "the worst pain imaginable").
Degree of patient satisfaction | 24 hours postoperatively
  The degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
Incidence of Complications | 24 hours postoperatively
  Incidence of complications as local anesthetic systemic toxicity, nerve injury, diaphragmatic paresis, pneumothorax and high epidural block.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.